CLINICAL TRIAL: NCT06758245
Title: Comparison of Anesthetic and Postoperative Analgesic Efficacy of Femoral and Popliteal Sciatic Block Application With Femoral and Anterior Sciatic Block Application in Ankle Surgery
Brief Title: Comparative Efficacy of Sciatic and Femoral Blocks in Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, principal investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GAZİOSMANPASATREHTAa
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain Management; Postoperative Pain; Analgesia; Nerve Blocks; Ankle Surgery
Keywords: nerve blocks; ankle surgery; postoperative pain; sciatic block; femoral block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral-Anterior sciatic block group (Active Comparator): First, in the supine position, the USG probe is placed below the inguinal crease. The femoral nerve is located lateral to the femoral artery, above the iliopsoas muscle. Once the needle tip reaches the nerve, simultaneous nerve stimulation is applied. Patellar movement is observed due to quadriceps muscle contraction upon needle placement. After a negative aspiration test, 20 ml of local anesthetic is injected.For the anterior sciatic block, while the patient was in the supine position, a convex ultrasound (USG) probe was placed transversely approximately 10 cm distal to the inguinal ligament. After visualizing the sciatic nerve as a hyperechoic flat structure, the nerve stimulator was set to 1-1.5 mA, 0.1 ms, and 1 Hz. Using an in-plane technique, the block needle was advanced. Upon reaching the sciatic nerve, when contractions in the calf, foot, or big toe continued at a current of 0.3-0.5 mA, 20 ml of 0.5% bupivacaine was administered following a negative aspiration test.
  Interventions: Procedure: femoral and anterior sciatic nerve block
- Femoral-popliteal sciatic block group (Active Comparator): First, in the supine position, the USG probe is placed below the inguinal crease. The femoral nerve is located lateral to the femoral artery, above the iliopsoas muscle. Once the needle tip reaches the nerve, simultaneous nerve stimulation is applied. Patellar movement is observed due to quadriceps muscle contraction upon needle placement. After a negative aspiration test, 20 ml of local anesthetic is injected.The ultrasound probe is placed transversely at the popliteal crease. The first structure seen is the popliteal artery. Just above and lateral to the artery, the tibial nerve appears as a hyperechoic, oval, and round structure. After identifying the tibial and peroneal nerves, the probe is moved proximally, and it is observed that the nerves join about 5-10 cm above the popliteal crease. The needle is advanced using an in-plane technique. After obtaining the first sciatic nerve stimulation, 20 cc of 0.5% bupivacaine is injected following a negative aspiration test.
  Interventions: Procedure: femoral and popliteal sciatic nerve block

INTERVENTIONS:
Procedure: femoral and anterior sciatic nerve block — First, in the supine position, the USG probe is placed below the inguinal crease. The femoral nerve is located lateral to the femoral artery, above the iliopsoas muscle. Once the needle tip reaches the nerve, simultaneous nerve stimulation is applied. Patellar movement is observed due to quadriceps muscle contraction upon needle placement. After a negative aspiration test, 20 ml of local anesthetic is injected.For the anterior sciatic block, while the patient was in the supine position, a convex ultrasound (USG) probe was placed transversely approximately 10 cm distal to the inguinal ligament. After visualizing the sciatic nerve as a hyperechoic flat structure, the nerve stimulator was set to 1-1.5 mA, 0.1 ms, and 1 Hz. Using an in-plane technique, the block needle was advanced. Upon reaching the sciatic nerve, when contractions in the calf, foot, or big toe continued at a current of 0.3-0.5 mA, 20 ml of 0.5% bupivacaine was administered following a negative aspiration test.
  Arms: Femoral-Anterior sciatic block group
Procedure: femoral and popliteal sciatic nerve block — The ultrasound probe is placed transversely at the popliteal crease. The first structure seen is the popliteal artery. Just above and lateral to the artery, the tibial nerve appears as a hyperechoic, oval, and round structure. After identifying the tibial and peroneal nerves, the probe is moved proximally, and it is observed that the nerves join about 5-10 cm above the popliteal crease. The needle is advanced using an in-plane technique. After obtaining the first sciatic nerve stimulation, 20 cc of 0.5% bupivacaine is injected following a negative aspiration test.
  Arms: Femoral-popliteal sciatic block group

SUMMARY:
Comparison of Anesthetic and Postoperative Analgesic Efficacy of Femoral and Popliteal Sciatic Block vs Femoral and Anterior Sciatic Block in Ankle Surgery

DETAILED DESCRIPTION:
The sciatic nerve, which arises from the sacral plexus, is the largest nerve in the body. It originates in the posterior region of the thigh in the lumbosacral area and is formed from the anterior branches of spinal nerves from L4 to S3 within the pelvis. It exits the pelvis through the greater sciatic foramen directly below the piriformis and then progresses towards the posterior compartment of the thigh, where it usually divides into the common peroneal nerve and the tibial nerve at the upper corner of the popliteal fossa. Sciatic nerve blocks provide both analgesia and anesthesia in surgeries below the knee, knee surgeries involving the posterior compartment, and foot and ankle surgeries. They can be used alone or in combination with an ipsilateral lumbar plexus block or femoral nerve block to provide surgical anesthesia or analgesia for the entire lower extremity.

Various approaches have been described to perform sciatic nerve block, including anterior and popliteal approaches. The anterior approach to the sciatic nerve can be performed as easily and successfully under ultrasound guidance as the popliteal approach. The anterior approach is advantageous when combined with a femoral nerve block, as it is performed with the patient in the supine position. Due to ease of application and high success rates, peripheral blocks have begun to be incorporated into anesthesia and postoperative analgesia strategies in ankle surgeries. The use of ultrasonography plays a crucial role in increasing the success rate of the block and reducing potential complications.

ELIGIBILITY:
* Inclusion Criteria:
* 18-65 years of age
* American Society of Anesthesiologists physical statusⅠ-II

Exclusion Criteria:

* Pregnant
* Neuromuscular disease
* Peripheral neuropathy
* Coagulation disorders
* Allergy to local anesthetics
* Infection at the site where the nerve block will be applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale values | at 1st, 4th,8th 12th ,24th and 48th hours after the surgery
  Visual Analogue Scale is a scale of 0-10 cm in length, expressed by non-standard verbal descriptors (no pain-unbearable pain..) indicating the limits of pain intensity on both sides, horizontally or vertically.

SECONDARY OUTCOMES:
Total amount of opioid requirements | within 48 hours after the surgery
  The total tramadol use of the patients in 48 hours will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Döndü GENÇ MORALAR, MD, Principal Investigator — GAZİOSMANPAŞA RESEARCH AND TRAİNİNG HOSPİTAL
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpasa Training and Research Hospital, Istanbul, 34000, Istanbul, Gaziosmanpasa
  - Gaziosmanpasa Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Olofsson M, Nguyen A, Rossel JB, Albrecht E. Duration of analgesia after forefoot surgery compared between an ankle and a sciatic nerve block at the popliteal crease: A randomised controlled single-blinded trial. Eur J Anaesthesiol. 2024 Jan 1;41(1):55-60. doi: 10.1097/EJA.0000000000001929. Epub 2023 Nov 16. PMID 37972929